CLINICAL TRIAL: NCT07066410
Title: Evaluation of the Effect of Different Calcium Silicate Cements on the Success of Vital Pulp Therapy in Irreversible Pulpal Infection Cases With Mature Roots: A Randomized Clinical Trial
Brief Title: Evaluation of Two Different Calcium Silicate Cements as a Treatment for Irreversible Pulpitis in Mature Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Yassmin, Yasmeen El-shaarawi, BDS, MSc Candidate, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-047
Record Dates: First submitted 2025-06-30; First posted 2025-07-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Irreversible Pulpitis
Keywords: Vital pulp therapy; Biodentine; Endocem; Irreversible pulpitis; MTA Pulpotomy; Pulpotomy in mature teeth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm 1 Endocem group (Experimental): Biological/Vaccine:
  Patients will undergo pulpotomy using EndoCem (Maruchi, Korea) after achieving hemostasis. Same standardized clinical procedure as the Biodentine group, but with EndoCem material used for pulp capping and final restoration placement.
  Interventions: Biological: intervention 1: endocem
- arm 2: Biodentine (Active Comparator): Patients will undergo pulpotomy using Biodentine (Septodont, France) after achieving hemostasis. Standardized clinical procedure including anesthesia, rubber dam isolation, access cavity preparation, coronal pulp removal, and placement of Biodentine followed
  Interventions: Biological: Intervention 1: biodentine

INTERVENTIONS:
Biological: intervention 1: endocem — EndoCem, a premixed calcium silicate-based cement (Maruchi, Korea), is used as the pulp capping material in vital pulp therapy (VPT). After achieving hemostasis with sterile saline-soaked cotton pellets, EndoCem is applied directly over the exposed radicular pulp tissue. The standardized clinical procedure includes local anesthesia, rubber dam isolation, caries removal, access cavity preparation, coronal pulp removal, and placement of EndoCem, followed by immediate restoration with FUJI II ensure a coronal seal.
  Arms: arm 1 Endocem group
Biological: Intervention 1: biodentine — Biodentine, a tricalcium silicate-based cement (Septodont, France), is used as the pulp capping material in vital pulp therapy (VPT). After achieving hemostasis with sterile saline-soaked cotton pellets, Biodentine is applied directly over the exposed radicular pulp tissue. The standardized clinical procedure includes local anesthesia, rubber dam isolation, caries removal, access cavity preparation, coronal pulp removal, and placement of Biodentine, followed by immediate restoration with FUJI II to ensure a coronal seal.
  Arms: arm 2: Biodentine

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of two calcium silicate cements-Biodentine and EndoCem-on post-operative pain and treatment success in vital pulp therapy (VPT) for mature permanent mandibular molars diagnosed with irreversible pulpitis. A total of 50 patients will be randomly assigned into two groups to receive pulpotomy using either Biodentine or EndoCem. The trial is triple-blinded, self-funded, and conducted at the Endodontic Department, Faculty of Dentistry, The British University in Egypt.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the impact of Biodentine and EndoCem on post-operative pain and treatment success in vital pulp therapy (VPT) of mature permanent mandibular molars with symptomatic irreversible pulpitis.

VPT preserves the vitality of radicular pulp by removing inflamed coronal pulp tissue and capping the remaining healthy pulp with a biocompatible material. This conservative approach may maintain pulp vitality, reduce treatment time, and improve patient outcomes compared to conventional root canal treatment.

Fifty eligible patients will be randomly assigned into two groups (n=25 per group). Pulpotomy will be performed under rubber dam isolation. After caries removal and coronal pulp amputation, hemostasis will be attempted with sterile saline-soaked cotton pellets. If bleeding persists beyond 5 minutes, the tooth will be excluded. The remaining pulp tissue will be capped with either Biodentine (Group 1) or EndoCem (Group 2), followed by immediate permanent restoration with composite resin to ensure a coronal seal.

Eligibility Criteria

Inclusion Criteria:

* Patients aged 12-40 years.
* Two-rooted mandibular molars diagnosed with symptomatic irreversible pulpitis.
* Restorable teeth.
* Periodontally healthy teeth (no mobility; negative percussion and palpation).
* Ability to provide informed consent.

Exclusion Criteria:

* Teeth with immature roots.
* Non-restorable teeth.
* Uncontrolled bleeding from the pulp after pulpotomy for more than 10 minutes.
* Necrotic teeth.
* Medically compromised patients with systemic conditions affecting treatment.
* Patients unable to provide informed consent.
* Vulnerable populations (e.g., minors without guardian consent).

Outcome Measures

Primary Outcome:

* Post-operative pain assessed using a Visual Analogue Scale (VAS; range 0-10, where 0 = no pain and 10 = worst possible pain). Time points: 6, 24, 48, and 72 hours post-treatment.

Secondary Outcome:

* Treatment success evaluated clinically (absence of pain, swelling, sinus tract) and radiographically (absence of periapical pathology) at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • Patient's age ranges from 12-40 years old.

  * Two Rooted Mandibular Molar teeth diagnosed with symptomatic irreversible pulpitis
  * The teeth are restorable
  * Informed consent granted
  * Teeth are periodontally free, with no mobility and negative to percussion and palpation test.

Exclusion Criteria:

* Teeth with immature roots

  * Non restorable teeth
  * Bleeding could not be controlled after pulpotomy in 10 minutes
  * Medically compromised patients with systemic complication that would alter the treatment.
  * Necrotic teeth
  * Inability to give informed consent

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Time Frame: at 6 hours, 24 hours, 48 hours, and 72 hours after treatment
  Pain intensity measured using the Visual Analogue Scale (VAS), a 100 mm scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate worse pain

SECONDARY OUTCOMES:
Success Rate | follow up at 3 and 6 months
  Teeth will be evaluated clinically for any signs or symptoms of pathosis including pain swelling sinus tract formation mobility and probing depth. teeth will be radiographically evaluated under optimum conditions, searching for periradicular pathosis, root resorption or internal resorption.Case will be considered successful if no clinical signs or symptoms and no radiographic sign of pathosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic at the British University in Egypt Hospital, Cairo, Cairo Governorate, Egypt